CLINICAL TRIAL: NCT01207518
Title: Cluster RCT Evaluating the Effectiveness of "Successful Influenza Immunization Campaigns in Healthcare Organizations: A Guide for Campaign Planners, Part of Optimizing Healthcare Workers Interpandemic Vaccine Uptake Study
Brief Title: Cluster RCT - Evaluating Effectiveness of a Guide and Tools for Influenza Immunization Campaign Planners
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Bruyère Health Research Institute. (Other); Canadian Center for Vaccinology (Other)
Responsible Party: Anne McCarthy, Ottawa Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Guide Cluster RCT
Record Dates: First submitted 2010-09-21; First posted 2010-09-23 (Estimated); Last update posted 2011-07-28 (Estimated); Status verified 2011-07

CONDITIONS: Influenza
Keywords: influenza; immunization; healthcare personnel
MeSH Terms: conditions — Influenza, Human | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): For the intervention group, there will be a Guide facilitator provided by the project team, normally the Project Manager or their delegate. The role of the Guide facilitator will be to provide basic information about the Guide and to facilitate the use of the web-based tools.
  Interventions: Behavioral: Intervention Group
- Control Group (Active Comparator): The Control Group will be asked to provide immunization rates for the base year and two years of the study, and will be asked about their influenza immunization campaign activities to use as a comparator. They will receive the Guide and web-based tools following completion of the study.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Intervention Group — This group of healthcare organizations will be given the Guide, web-based tools and access to a Guide facilitator throughout the study.
  Arms: Intervention Group
Behavioral: Control Group — This group will provide their immunization rates for the base and study years and will provide information on their campaign activities. No other intervention will be provided.
  Arms: Control Group

SUMMARY:
During the 2010-2011 and the 2011-2012 seasonal influenza immunization campaigns, we will recruit a minimum of 46 healthcare organizations to either conduct their campaigns as usual or to use the "Successful Influenza Immunization Campaigns for Healthcare Personnel: A Guide for Campaign Planners and a web-based grab-and-go Tool Kit. At the end of the campaign season we will evaluate the impact of the Guide and web-based tools and assess whether there were changes in immunization rates within each organization and/or if there were significant changes in the management of the campaigns across organizations.

Following completion of the study, we will work with partner organizations to make these tools available to all Canadian healthcare organizations.

DETAILED DESCRIPTION:
Keeping nurses, physicians and allied health professionals working during seasonal influenza epidemics is essential. Influenza immunization has been shown to mitigate the adverse health outcomes associated with influenza in the community. When provided to healthcare personnel, influenza vaccine reduces the frequency and severity of influenza outbreaks and reduces influenza-associated morbidity and mortality among patients by reducing the transmission of influenza from healthcare personnel to their vulnerable patients.

Despite abundant evidence of the safety and efficacy of the influenza vaccine, immunization rates among healthcare personnel in hospital and long-term settings remain well below the public health target of 90%. Current initiatives targeted at increasing healthcare personnel immunization rates are having limited success with healthcare personnel immunization rates as low as 2%, but averaging 40% - 60% in most healthcare facilities being reported.

Following the work of the research team over the past two years, a Guide, called "Successful Influenza Immunization Campaigns for Healthcare Personnel: A Guide for Campaign Planners" has been developed, along with web-based "grab and go" tools (the Toolkit). This practical Guide is structured to facilitate the use of the evidence-based research on strategies to increase immunization rates by healthcare planners.

ELIGIBILITY:
Inclusion Criteria:

At least 46 healthcare organizations from across Canada will be selected to participate in the study.

The Guide is designed to be used across different types of healthcare organizations. Potential healthcare organizations will be self-identified, recommended by a project team member, and/or selected from the Canadian Healthcare Association's Guide to Healthcare Facilities. Selected sites must meet the following eligibility criteria:

* Canadian healthcare organizations who conduct seasonal influenza immunization campaigns
* Have a systematic approach to collecting healthcare personnel immunization rates and be able to provide accurate and timely reports of immunization rates for categories of healthcare personnel
* Agree to be randomized to receive the Guide or receive no intervention
* If randomized to receive the Guide, the organization, including the campaign team and senior management, agrees to commit to adhere to the steps in the Guide to plan, implement, monitor and evaluate their campaign

Exclusion Criteria:

Healthcare organizations who do not meet the above criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-03 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Intervention Group - 10% improvement in immunization rates | 2010 to 2012
  In the Intervention Group, a 10% improvement in healthcare personnel immunization rates from the base year (2008-2009) as compared to Year One (2010-2011) and Year Two (2011-2012), assessed using a time-series analysis on how each organization does against themselves and between the Intervention and Control Group. We will also the WHO benchmark of 90%.

SECONDARY OUTCOMES:
Improvement in the reporting of immunization rates | 2010-2012
  In both the Intervention and Control Group, we will assess improvement in the reporting of immunization rates, based on the methodology outlined in Appendix 3 of the Guide.

CONTACTS AND LOCATIONS:
Overall Officials: Larry W Chambers, PhD(Epi), Principal Investigator — Bruyère Health Research Institute.
Locations (2):
- Canada (2):
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Élisabeth Bruyère Research Institute, Ottawa, Ontario

REFERENCES:
- [Background] Lam PP, Chambers LW, MacDougall DM, McCarthy AE. Seasonal influenza vaccination campaigns for health care personnel: systematic review. CMAJ. 2010 Sep 7;182(12):E542-8. doi: 10.1503/cmaj.091304. Epub 2010 Jul 19. PMID 20643836
- [Derived] Chambers LW, Crowe L, Lam PP, MacDougall D, McNeil S, Roth V, Suh K, Dalzell C, Baker D, Ramsay H, DeCoutere S, Hall HL, McCarthy AE. A new approach to improving healthcare personnel influenza immunization programs: a randomized controlled trial. PLoS One. 2015 Mar 17;10(3):e0118368. doi: 10.1371/journal.pone.0118368. eCollection 2015. PMID 25781888